CLINICAL TRIAL: NCT05973383
Title: Effectiveness and Theory-based Evaluation of a Personalised Digital Intervention (EviBody) for Healthy and Sustained Lifestyle Behaviours and Well-being Among Adults
Brief Title: Evaluation of a Personalised Digital Intervention (EviBody) for Healthy and Sustained Lifestyle Behaviors and Well-being Among Adults: a Real-world Quasi-experimental Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sophiahemmet University (Other)
Collaborators: Karolinska Institutet (Other); Stockholm University (Other); The Swedish School of Sport and Health Sciences (Other); Linnaeus University (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-23-07-043416
Record Dates: First submitted 2023-07-08; First posted 2023-08-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Well-being
Keywords: primary prevention; secondary prevention; health promotion; self-management; behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intervention group- Basic: Subjects with behavioral support from the app EviBody
  Interventions: Behavioral: EviBody- Basic
- Intervention group- Standard: Subjects with behavioral support from the app EviBody + social support
  Interventions: Behavioral: EviBody- Standard
- Intervention group- Premium: Subjects with behavioral support from the app EviBody + social support + individual coaching
  Interventions: Behavioral: EviBody- Premium
- Control group: No exposure

INTERVENTIONS:
Behavioral: EviBody- Basic — The app EviBody with three core subjects:
  1) a Healthy eating, 2) Physical activity, and 3) Mental balance. The intervention includes tracking and self-monitoring of behaviors, goal setting, action planning, feedback and digital rewards, an AI chat, a database with food recipes, a database with exercises, inspiration, and skills training webinars.
  Groups: Intervention group- Basic
Behavioral: EviBody- Standard — The digital service EviBody with three core subjects:
  1) a Healthy diet, 2) Physical activity, and 3) Mental balance. The service includes tracking and self-monitoring of behaviors, goal setting, action planning, feedback and digital rewards, an AI chat, a database with food recipes, a database with exercises, inspiration, and skills training webinars.
  Users with the membership Standard are also offered a community with social support.
  Groups: Intervention group- Standard
Behavioral: EviBody- Premium — The digital service EviBody with three core subjects:
  1) a Healthy diet, 2) Physical activity, and 3) Mental balance. The service includes tracking and self-monitoring of behaviors, goal setting, action planning, feedback and digital rewards, an AI chat, a database with food recipes, a database with exercises, inspiration, and skills training webinars.
  Users with the membership Premium are also offered a community with social support plus private on-line health consultations. The number of private health consultations is 3 for a 3 months subscription, 4 for a 6 months subscription, and 6 for a 12 months subscription.
  Groups: Intervention group- Premium

SUMMARY:
The goal of this quasi-experimental observational study is to evaluate the impact of a personally tailored digital intervention aimed to support a healthy lifestyle on well-being, lifestyle behaviors, and mental health among the adult population.

The main questions it aims to answer are:

I) Is a digital intervention developed to offer personalised digital support for healthy habits effective in improving well-being compared to a control group from the general population after 6 months? II) Is the effectiveness dose-dependent (better effect with higher membership level)? III) Does the digital intervention assist in maintaining healthy eating and physical activity habits, mental health, and well-being across 24 months? IV) Are sociodemographic factors associated with achieving the self-identified goals and improvements in eating and physical activity habits, mental health, and well-being? VI) Do engagement, motivation, self-efficacy, and perceived barriers mediate the associations between sociodemographic characteristics and changes in self-identified goals, eating and physical activity habits, mental health, and well-being over a 24-month period? V) How is the pattern of user engagement across 24 months?

Participants are users of the mobile phone application EviBody. The group will be compared with individuals from the general population to evaluate if the digital intervention is effective in improving well-being, eating and physical activity habits, and mental health.

DETAILED DESCRIPTION:
EviBody is a personally tailored digital intervention promoting healthy habits that is co-developed, based on behavioural research evidence, and supported by artificial intelligence.

The primary study is a quasi-experimental study with a non-randomised control group. A four-armed design will allow for comparison between three levels of intervention (basic, standard and premium) and a control group. The digital intervention (the app EviBody) will be marketed and managed by its owner LongLife Active AB (Limited Company), Sweden. Allocation to intervention arm is by preference (chosen membership level of the app) and takes place at enrolment. Being a research participant includes answering seven questionnaires during two years and allowing researchers to extract data from app analytics. Ethical approval was obtained from the Swedish Ethical Review Authority, Dnr 2023-06246-01 on January 30 2024.

ELIGIBILITY:
Inclusion Criteria (intervention arms):

* adults ≥18 years
* signing up for the app EviBody using electronic identification
* consent to the research study

Inclusion Criteria (controls):

* adults ≥18 years
* consent to the research study

Exclusion Criteria (intervention arms):

* individuals who are discharged from the app due to refracting the terms of the service,
* is currently using a digital product that is explicitly designed to support behaviour change,
* subjects scoring >70 on well-being will be excluded from the primary analyses,
* subjects who appear as friends, colleagues, or family with anyone in the research or owner group will be excluded.

Exclusion Criteria (controls):

* is currently using a digital product that is explicitly designed to support behaviour change,
* is found to be a user of EviBody,
* subjects scoring >70 on well-being will be excluded from the primary analyses,
* subjects who appear as friends, colleagues, or family with anyone in the research or owner group will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intervention:
  Adults signing up for a digital intervention that is supporting a healthy lifestyle.
  Control:
  Adults of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Well-being | 6 months
  Well-being will be assessed by the WHO-5 Well-Being Index. The WHO-5 comprises the following five items: being cheerful and in good spirits; being calm and relaxed; feeling active and vigorous; feeling fresh and rested when waking up in the morning; and having an interest in day-to-day activities. Six response alternatives are scored from 5 (All of the time) to 0 (At no time). The total raw score which ranges from 0 to 25 is multiplied by 4 to calculate the final score. The final score range goes from 0 = worst imaginable well-being to 100 = the best imaginable well-being.
Well-being | 24 months
  Well-being will be assessed by the WHO-5 Well-Being Index. The WHO-5 comprises the following five items: being cheerful and in good spirits; being calm and relaxed; feeling active and vigorous; feeling fresh and rested when waking up in the morning; and having an interest in day-to-day activities. Six response alternatives are scored from 5 (All of the time) to 0 (At no time). The total raw score which ranges from 0 to 25 is multiplied by 4 to calculate the final score. The final score range goes from 0 = worst imaginable well-being to 100 = the best imaginable well-being.

SECONDARY OUTCOMES:
Stress | 6 months
  Stress will be assessed by the Karolinska Exhaustion Disorder Scale (KEDS), a self-rating scale for stress-induced exhaustion disorder. 9 items are scored 1-6, a higher total score indicates more exhaustion.
Burnout | 6 months
  Burnout will be assessed by the Oldenburg Burnout Inventory (OLBI). 16 items are scored 1-4, a higher total score indicates more burnout.
Sleep | 6 months
  Sleep will be assessed by the self-reported number of hours of sleep per night and by Insomnia Severity Index (ISI). In ISI 7 items are scored 1-4 and a higher total score indicates more sleeping problems.
Stress | 24 months
  Stress will be assessed by the Karolinska Exhaustion Disorder Scale (KEDS), a self-rating scale for stress-induced exhaustion disorder. 9 items are scored 1-6, a higher total score indicates more exhaustion.
Burnout | 24 months
  Burnout will be assessed by the Oldenburg Burnout Inventory (OLBI). 16 items are scored 1-4, a higher total score indicates more burnout.
Sleep | 24 months
  Sleep will be assessed by the self-reported number of hours of sleep per night and by Insomnia Severity Index (ISI). In ISI 7 items are scored 1-4 and a higher total score indicates more sleeping problems.

OTHER OUTCOMES:
Goal achievement | 6 months
  Reaching the self-identified goal will be evaluated by collecting information on number of days/week the self-identified goal was met during the past month. Confidence for reaching the goal will also be asked for on a scale 1 low confidence to 6 high confidence.
Dietary habits | 6 months
  Dietary behaviours will be assessed by questions from the Social Board of Health and Welfare in Sweden, with the addition of some study specific questions on plant based diet.
Physical activity | 6 months
  Physical activity will be collected by questions from the Social Board of Health and Welfare with additional questions on active transport and physical activity at work. In a randomized sample of individuals having increased physical activity as a goal (n=300) physical activity will also be measured objectively by the use of the three-axial accelerometer-based device.
Sedentary behavior | 6 months
  Sedentary behavior will be collected by questions from the Social Board of Health and Welfare with additional questions on active transport and physical activity at work. In a randomized sample of individuals having increased physical activity as a goal (n=300) physical activity will also be measured objectively by the use of the three-axial accelerometer-based device.
Daily number of steps | 6 months
  Daily number of steps will be obtained from app analytics.
Goal achievement | 24 months
  Reaching the self-identified goal will be evaluated by collecting information on number of days/week the self-identified goal was met during the past month. Confidence for reaching the goal will also be asked for on a scale 1 low confidence to 6 high confidence.
Dietary habits | 24 months
  Dietary behaviours will be assessed by questions from the Social Board of Health and Welfare in Sweden, with the addition of some study specific questions on plant based diet.
Physical activity | 24 months
  Physical activity will be collected by questions from the Social Board of Health and Welfare with additional questions on active transport and physical activity at work. In a randomized sample of individuals having increased physical activity as a goal (n=300) physical activity will also be measured objectively by the use of the three-axial accelerometer-based device.
Sedentary behavior | 24 months
  Sedentary behavior will be collected by questions from the Social Board of Health and Welfare with additional questions on active transport and physical activity at work. In a randomized sample of individuals having increased physical activity as a goal (n=300) physical activity will also be measured objectively by the use of the three-axial accelerometer-based device.
Daily number of steps | 24 months
  Daily number of steps will be obtained from app analytics.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Rossen, PhD, Principal Investigator — Sophiahemmet University

REFERENCES:
- [Derived] Rossen J, Anderbro T, Andermo S, Bergman P, Hagstromer M, Jacobsson M, Johansson UB, Kallings L, Lonn A, Regan C, von Rosen P. Effectiveness and theory-based evaluation of a personalised digital intervention (EviBody(R)) for healthy and sustained lifestyle behaviours and well-being among adults: Study protocol for a real-world quasi-experimental study. PLoS One. 2025 Oct 7;20(10):e0333201. doi: 10.1371/journal.pone.0333201. eCollection 2025. PMID 41056320
- See also: Research project website — https://www.shh.se/en/research-fields/longlife-active-an-individually-tailored-digital-service-to-promote-healthy-and-sustainable-behaviors-supported-by-ai/